CLINICAL TRIAL: NCT00928551
Title: A Randomized, Open-Label, Single-Dose, 3-Period Crossover, Comparative Study of a Modified Formulation of Vabicaserin (SCA-136) Versus the Reference Formulation in Healthy Subjects
Brief Title: Comparative Formulation Study of Vabicaserin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3153B3-1128
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — vabicaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: vabicaserin

INTERVENTIONS:
Drug: vabicaserin

SUMMARY:
This study will compare two different formulations of vabicaserin.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after investigational product administration.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion Criteria:

* Use of any investigational or prescription drug within 30 days before investigation product administration.
* Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before study day 1.
* Use of any over-the-counter drugs, including herbal supplements within 72 hours before study day 1.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters including plasma concentrations, Cmax, and AUC. | 2 months

SECONDARY OUTCOMES:
Safety assessment as measured by evaluating any reported adverse events, scheduled physical examinations, vital sign measurements, ECGs, and clinical laboratory results. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Brighton, Massachusetts, United States